CLINICAL TRIAL: NCT07135778
Title: The Efficacy and Safety of Liposomal Amphotericin B and Isavuconazole/Posaconazole in the Treatment of Breakthrough Invasive Fungal Disease in Patients With Malignant Hematological Diseases After Antifungal Prophylaxis
Brief Title: Liposomal Amphotericin B and Isavuconazole/Posaconazole in Br-IFD（ Breakthrough Invasive Fungal Disease） in Patients With Malignant Hematological Diseases
Status: Recruiting | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QTJC2025031
Record Dates: First submitted 2025-07-31; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-06

CONDITIONS: Invasive Fungal Disease
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Non-Probability Sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: patients received L-AmB therapy: Dose: 3-5mg/kg/day administered intravenouly(IV). Duration of treatment: Researchers determine based on the severity of the underlying disease, the recovery of immune suppression, and clinical response.
  All drug dosages are in accordance with the drug instructions.All treatments must be prescribed according to local routine clinical practice, and the preparation and administration of drugs must be carried out in accordance with the instructions and guidelines provided by the manufacturer.
- Group 2: patients received isavuconazole/posaconzazole therapy: Foumulations: Oral tablets or intravenous (IV) formulations. Dosing: Loading dose: As per product labeling. Maintenance dose: 300mg (posaconzazole) or 200mg (isavuconazole) once daily. Duration of treatment: Researchers determine based on the severity of the underlying disease, the recovery of immune suppression, and clinical response.
  All drug dosages are in accordance with the drug instructions. All treatments must be prescribed according to local routine clinical practice, and the preparation and administration of drugs must be carried out in accordance with the instructions and guidelines provided by the manufacturer.

SUMMARY:
This is a prospective, open label, controlled, single center real-world observational study. Adult (aged ≥ 18 years) patients with hematological malignancies develop breakthrough invasive fungal disease after receiving ≥ 7 days of echinocandin or triazole antifungal prophylaxis receive treatment with liposomal amphotericin B or treatment with Isavuconazole or posaconazole according to the clinical doctor's decision. It is planed to collect 36 patients receiving treatment with liposomal amphotericin B and 36 patients receiving treatment with Isavuconazole or posaconazole, and observe their efficacy and safety.

DETAILED DESCRIPTION:
This is a prospective, open label, controlled, single center real-world observational study. Adult (aged ≥ 18 years) patients with hematological malignancies develop breakthrough invasive fungal disease after receiving ≥ 7 days of echinocandin or triazole antifungal prophylaxis receive treatment with liposomal amphotericin B or treatment with Isavuconazole or posaconazole according to the clinical doctor's decision. It is planed to collect 36 patients receiving treatment with liposomal amphotericin B and 36 patients receiving treatment with Isavuconazole or posaconazole, and observe their efficacy and safety. The research objective of this study is to: 1. Evaluate efficacy: The main objective is to determine the therapeutic effect of L-AmB (liposomal amphotericin B) or Isavuconazole/posaconazole on breakthrough invasive fungal disease, including percentage of patients with favorable overall response, survival rate, median to fever remission time, length of hospital stay, etc.2. Evaluate safety: Study the safety of drugs, including monitoring and recording all adverse events, side effects, and drug-related toxicity. 3. Patient population analysis: Study the differences in response to treatment with liposomal amphotericin B and Isavuconazole/posaconazole among different patient populations (such as different ages, genders, and underlying disease states).

These research objectives will contribute to a comprehensive understanding of the roles of L-AmB and Isavuconazole/posaconazole in the treatment of breakthrough fungal infections, and provide scientific evidence for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged ≥ 18 years at the beginning of treatment.
* The patient or their guardian must be able to understand and sign a written informed consent form (which must be obtained before starting any research procedure)
* Blood based diseases, mainly AML( Acute Myeloid Leukemia), ALL(Acute Lymphoblastic Leukemia), MDS(Myelodysplastic Syndromes)
* Breakthrough invasive fungal disease occurs after receiving antifungal prophylaxis with triazole drugs for ≥ 7 days
* According to the latest definition of MSGERC, breakthrough IFD is defined as any IFD that occurs during exposure to antifungal drugs, including fungal infections outside the spectrum of antifungal activity
* Proven, probable, and possible IFD in accordance with the< The Chinese guidelines for the diagnosis and treatment of invasive fungal disease in patients with hematological disorders and cancers (the 6th revision) >

Exclusion Criteria:

* Confirmed patients with allergies/rapid onset severe allergic reactions/intolerance to L-AmB or isavuconazole /posaconazole
* Serum creatinine level ≥ 2 times the upper limit of normal
* The level of transaminase or alkaline phosphatase is ≥ 5 times the normal upper limit, and bilirubin is ≥ 3 times the normal upper limit
* Patients who are breastfeeding
* Pregnant patients
* Expected life expectancy is less than 30 days
* Patients deemed ineligible by the investigator due to medical, ethical, or logistical reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breakthrough invasive fungal disease in patients with malignant hematological diseases after antifungal prophylaxis
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The favorable overall responses rate at the end of treatment (proportion of patients achieving complete or partial remission) | through study completion, an average of 2 weeks
  The end of treatment refers to the time when L-AmB or Isavuconazole/posaconazole treatment ends.
  According to the EORTC/MSG (European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group and the National Institute of Allergy and Infectious Diseases Mycosis Study Group)efficacy evaluation criteria based on clinical evaluation, the response is divided into complete remission, partial remission, disease stability, disease progression, and death directly related to the study drug or IFD(invasive fungal disease). Effective refers to complete and partial remission.

SECONDARY OUTCOMES:
Survival rate at key time points | through study completion, an average of 2 weeks
  proportion of participants alive at (1) end of treatment (2) 42 days post-therapy (3)84 days post-therapy. Survival is defined as being free from death due to any cause
Time to favorable overall response | 14 days
  Duration from study enrollment to achievement of a favorable overall response (complete or partial resolution of mucormycosis symptoms, radiological improvement, and microbiological clearance)
Length of hospitalization | 30 days
  Total number of days participants spend hospitalized from enrollment until discharge or death.
incidence of treatment-emergent adverse events | 30 days
  incidence and severity of treatment-emergent adverse events(TEAEs), including nephrotoxicity, hepatotoxicity, infusion reactions, and electrolyte abnormalities, graded per CTCAE V5.0(National Cancer Institute - Common Terminology Criteria for Adverse Events Version 5.0) criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- National Clinical Research Center for Blood Diseases, Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD